CLINICAL TRIAL: NCT01756911
Title: Evaluation du Stent Multicouches Dans le Traitement Des anévrismes de l'Aorte Thoraco-abdominale
Brief Title: Evaluation of the Safety and Efficacy of the Multilayer Stent
Acronym: STRATO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiatis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC_0308_FRA; 2009-013678-42 (EudraCT Number)
Record Dates: First submitted 2012-12-14; First posted 2012-12-28 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Aortic Aneurysm, Thoracoabdominal; Thoracoabdominal Aortic Aneurysm; Aortic Aneurysm, Thoracic
Keywords: MFM; Multilayer Flow Modulator; Multilayer stent; Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thotaco-abdominal aneurysm (Experimental): MFM
  Interventions: Device: MFM

INTERVENTIONS:
Device: MFM — Implantation of the MFM
  Other Names: Multilayer Flow Modulator; Multilayer stent

SUMMARY:
Evaluation of the Multilayer Flow Modulator (MFM) for Endovascular Thoracoabdominal Aneurysm Repair.

The objectives of the study is to determine the efficacy, safety and performance of the MFM and its delivery system in patients at high surgical risk presenting with a type II, III thoracoabdominal aneurysm, below the left subclavian and above the iliac bifurcation, according to the Crawford classification.

DETAILED DESCRIPTION:
Conventional treatments of thoracoabdominal aneurysm are medical treatments (based on hypertension control) on one hand and surgical treatment on the other hand.

The standard treatment is surgery consisting of an exclusion of the aneurysm with restoration of continuity by means of a prosthesis usually made of Dacron.

* The rates of surgical morbidity and mortality differ according to whether the patient is treated electively or in an emergency setting. The most feared complication is spinal cord ischemia inducing paraplegia.
* In elective surgery, operative mortality is estimated to be between 6% and 15% depending on the series, and around 50% to 60% of patients are treated in an emergency setting. The rate of neurological complications such as paraparesis or paraplegia is estimated to be between 3% and 15%.
* In addition to the above, the following major complications have been shown to have an impact on the morbidity of this major surgery (5% each):
* Bleeding requiring surgical hemostasis
* Respiratory distress syndrome requiring prolonged ventilation support
* Acute renal failure
* Infections
* Central neurological events (stroke and coma)
* Peripheral neurological events (sensory-motor deficits, paraparesis, paraplegia)

Analyses identify risk factors increasing the morbidity and mortality:

* Patients over 80 years
* Chronic obstructive pulmonary disease
* Renal failure
* Coronary artery disease
* Comorbidities (malignancy, etc.)

Compared to surgery, endovascular stenting reduces:

* Pulmonary morbidity (suppression of thoracotomy and ventilation), in patients with impaired lung function;
* Renal dysfunction;
* Myocardial failure;
* Risk of spinal cord ischemia and paraplegia.

However, this treatment has a number of limitations

* Availability of device in case of emergency
* Topography of the neck must be far enough from the left subclavian artery to allow satisfactory fixation of the stent and exclusion of the lesion;
* Obstruction of the branches near the aneurysm.

In the current available treatment for this pathology, there are still some disadvantages such as the difficulty of precise positioning of the prosthesis and its branches which must cover the aneurysm tissue without endoleaks. Each lesion having anatomical specificities, the device must be designed for each individual patient, and the operator's technical ability must be extreme. So, the current technique is difficult to reproduce, and any emergency treatment is impossible.

The multilayer flow modulator (non-covered) is the device used in this trial The complications mentioned above are inherent in the concept of covered stent treatment plus endoleaks that continues to fuel the aneurismal sac untreated, thus subject to the persistent risk of rupture. With this technique, the visceral arteries are occluded or have a retrograde flow (which pressurizes the aneurysm again).

The multilayer flow modulator (non-covered) treatment approach avoids the major problems mentioned above:

* It allows the aneurismal sac to thrombose whilst maintaining the patency of collateral branches arising from the aneurysm;
* It improves the flow in the collateral branches, which becomes laminar flow through a mechanism of hemodynamic pressure drop from layer to layer and an increase in speed by rolling;
* Deployment is easier and it is not different from peripheral stent deployment;
* The device is available in all sizes and all lengths that can be stored, allowing the management of emergencies.

The space-age 3D geometrical design of a Cardiatis multilayer flow modulator modifies flow within the aorta in a way that reduces pressure within the aneurysm thus collapsing the aneurismal sac while preserving any vital collateral circulation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Life expectancy ≥ 12 months
* The patient or his legal representative has signed the informed consent form
* Thoracoabdominal aneurysm type 2 or 3 with vital collaterals and requiring intervention to prevent its rupture according to the criteria defined by consensus ("Expert Consensus Document on the Treatment of Descending Thoracic Aortic Disease Using Endovascular Stent-Grafts", Ann Thorac Surg 2008;85:S1-41)
* Contraindicated for open surgery, declared inoperable by the surgeon and anesthetist (statement signed by each doctor) and must have at least one of the following:

  1. Age > 80 years
  2. ASA (American Society of Anesthesiologists) score ≥ 3
  3. History of thoracic surgery or surgery of the abdominal aorta
  4. Coronary artery disease (history of angina or myocardial infarction) with positive functional testing and coronary lesions for which revascularization is impossible or not indicated
  5. Heart failure
  6. Inoperable aortic stenosis
  7. LVEF (Left Ventricular Ejection Fraction) <40%;
  8. chronic respiratory failure defined by one of the following criteria:

     1. FEV (Forced expiratory volume) <1.2 l / sec;
     2. VC (Vital Capacity) <50% of the predicted value according to age, sex and weight;
     3. arterial blood gas analysis in the absence of oxygen: PaCO2 (Pression artérielle en CO2) > 45 mmHg or PaO2 (Pression artérielle en O2) <60 mmHg
     4. Oxygen therapy
  9. renal insufficiency if creatininaemia> 200 micromol / l before injection of contrast product;
  10. hostile abdomen, including presence of ascites or other signs of portal hypertension;
  11. obesity.
* adequate arterial anatomy of aneurismal lesion access.

Exclusion Criteria:

* medical contraindications to a local or general anesthesia and angiography;
* Life expectancy less than one year, or clinical follow-up impossible;
* congenital disorders of blood coagulation;
* intercurrent infection;
* allergy to aspirin, clopidogrel, or contrast agents;
* patient(s) included in another clinical study;
* patient pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with aneurysm exclusion | 12 months

SECONDARY OUTCOMES:
Number of covered branches permeable | 12 months
Number of patients with Serious Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Noël Fabiani, Pr, Principal Investigator — HEGP
Locations (9):
- France (9):
  - Hopital Jean Minjoz, Besançon
  - Hopital Neurocardiologique, Bron
  - Centre Hospitalier de La Région D'Annecy, Metz-Tessy
  - Chu Brabois Nancy, Nancy
  - Hopital Europeen Georges-Pompidou, Paris
  - Pitie-Salpetriere, Paris
  - CMC Parly II, Paris
  - Institut Cardio-Vasculaire Paris Sud Hôpital Claude Galien À Quincy, Quincy-sous-Sénart
  - Hopital Universitaire Rangueil, Toulouse

REFERENCES:
- [Result] Vaislic CD, Fabiani JN, Chocron S, Robin J, Costache VS, Villemot JP, Alsac JM, Leprince PN, Unterseeh T, Portocarrero E, Glock Y, Rousseau H; STRATO Investigators Group. One-year outcomes following repair of thoracoabdominal aneurysms with the multilayer flow modulator: report from the STRATO trial. J Endovasc Ther. 2014 Feb;21(1):85-95. doi: 10.1583/13-4553R.1. PMID 24502488
- [Derived] Vaislic CD, Fabiani JN, Chocron S, Robin J, Costache VS, Villemot JP, Alsac JM, Leprince PN, Unterseeh T, Portocarrero E, Glock Y, Rousseau H; STRATO Investigators Group. Three-Year Outcomes With the Multilayer Flow Modulator for Repair of Thoracoabdominal Aneurysms: A Follow-up Report From the STRATO Trial. J Endovasc Ther. 2016 Oct;23(5):762-72. doi: 10.1177/1526602816653095. Epub 2016 Jun 8. PMID 27280802
- See also: One-year outcomes following repair of thoracoabdominal aneurysms with the multilayer flow modulator: report from the STRATO trial — http://www.ncbi.nlm.nih.gov/pubmed/24502488